CLINICAL TRIAL: NCT01876732
Title: Impact of Vitamin B12 Replacement on Epogen Dosing and Improvement of Quality of Life in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Nephrology Attending, Assoc. Chair of Medicine, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 09-024; NCT01360983 (obsolete NCT alias)
Record Dates: First submitted 2013-05-14; First posted 2013-06-13 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Vitamin B12 Deficiency
Keywords: hemodialysis; viatmin B12 deficiency; Epogen
MeSH Terms: conditions — Vitamin B 12 Deficiency | interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin B12 (Experimental): Those with an MMA over 800nmol/L are given 1000mcg of intramuscular (IM) vitamin B12 weekly for the first month and then monthly for 3 consecutive months.
  Interventions: Drug: Vitamin B12

INTERVENTIONS:
Drug: Vitamin B12 — Consented subjects are screened for Vitamin B12 deficiency with measurements of serum vitamin B12 concentrations and plasma levels of MMA, drawn prior to the first hemodialysis (HD) session of the week. Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months. Following therapy, serum B12, MMA levels, percent iron saturation, parathyroid levels and peripheral blood smear are to be repeated and compared to previous levels. Subjects also complete a Kidney Disease Quality of Life- 36 (KDQOL-36) prior to therapy and again post treatment.
  Other Names: Cyanocobalamin

SUMMARY:
Vitamin B12 has several important functions in the body, two of which are production of red blood cells and the maintenance of a healthy nervous system. When vitamin B12 is deficient, abnormal red blood cells form. These cells are called megaloblasts. The end result is a decreased number of red blood cells; a condition called anemia. Some symptoms of anemia include fatigue, weakness, shortness of breath, and pallor. Vitamin B12 is also important in maintaining a healthy nervous system. Nerves are surrounded by an insulating material that helps them conduct impulses. Patients with low B12 levels who receive this vitamin in injection form, state that there quality of life is better. Anemia in Hemodialysis patients is treated with Epogen, a synthetic material which helps your body make blood cells. The investigators believe that if you have a low vitamin B12 level in your blood and the investigators give you the vitamin during dialysis your requirement for epogen will be lower and you will be able to produce blood cells better. When evaluating for Vitamin B12 deficiency a special test is needed called methylmalonic acid level (MMA). This is a blood test that will be performed and when this level is high and your vitamin B12 level is in the low normal range the investigators can make a diagnosis of vitamin B12 deficiency.

DETAILED DESCRIPTION:
BACKGROUND: Vitamin B12 deficiency may have deleterious effects on end stage renal disease (ESRD) patients on maintenance hemodialysis, and may increase erythropoietin stimulating agent (ESA) resistance, yet little is known about its prevalence in this population.

METHODS: Serum vitamin B12 and methylmalonic acid (MMA) levels were drawn from ESRD patients prior to hemodialysis. All patients with MMA levels greater than 800 nmol/L had peripheral smears evaluated for B12 deficiency. Those with confirmatory smears were considered to be deficient and received intramuscular vitamin B12 injections for 4 months. Post-treatment MMA levels and smears were obtained. Erythropoietin dosages were monitored throughout the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* · Patients on Hemodialysis for at least 6 months

  * Patients on stable dose of epogen and iron supplementation for at least 1 month prior to B12 and MMA assay.

Exclusion Criteria:

* · On B12 treatment

  * Hematological Cancer
  * Methotrexate use
  * Alcohol use greater then 2 drinks per day
  * Vegetarian Diet
  * Gastric Surgery
  * Inflammatory Bowel Disease
  * Pernicious Anemia
  * Recent transfusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Principal Investigator — SIUH
Locations (1):
- Island Rehab, Staten Island, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months.
Groups:
- Vitamin B12: Those with an methylmalonic acid (MMA) over 800nmol/L are given 1000mcg of intramuscular (IM) vitamin B12 weekly for the first month and then monthly for 3 consecutive months.
  Vitamin B 12: Consented subjects are screened for Vitamin B12 deficiency with measurements of serum vitamin B12 concentrations and plasma levels of MMA, drawn prior to the first hemodialysis (HD) session of the week. Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months. Following therapy, serum B12, MMA levels, percent iron saturation, parathyroid levels and peripheral blood smear are to be repeated and compared to previous levels. Subjects also complete a Kidney Disease Quality of Life- 36 (KDQOL-36) prior to therapy and again post treatment.
Period: Overall Study
Arm/Group | Vitamin B12
Started | 132
Completed | 57
Not Completed | 75
Not completed — MMA was not over 800mg/dL | 75

BASELINE CHARACTERISTICS:
Groups:
- Vitamin B12: Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months.
Arm/Group | Vitamin B12
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants] — From a single center dialysis unit, patients 18-80 on hemodialysis at least 6 months and taking Epogen were screened for serum Vitamin B12 levels and plasma MMA. Those with an MMA level greater than 800mmol/L had smears of their peripheral blood examined to assess for characteristic findings that are consistent with vitamin B12 deficiency.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 50
    >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.43 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Primary Outcome: Change in Amount of Epogen Required
Description: The effects of Vitamin B12 supplementation on erythropoitin alpha (Epogen) requirements in HD patients
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: unit/ml
Groups:
- Vitamin B12: Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months.
  Vitamin B12: Consented subjects are screened for Vitamin B12 deficiency with measurements of serum vitamin B12 concentrations and plasma levels of MMA, drawn prior to the first HD session of the week. Those with an MMA over 800nmol/L are given 1000mcg of IM vitamin B12 weekly for the first month and then monthly for 3 consecutive months. Following therapy, serum B12, MMA levels, percent iron saturation, parathyroid levels and peripheral blood smear are to be repeated and compared to previous levels. Subjects also complete a KDQOL-36 prior to therapy and again post treatment.
Arm/Group | Vitamin B12
Number analyzed (Participants) | 57
unit/ml | -16,572 (41,902)

2. Secondary Outcome: Change in Quality of Life
Description: The scoring procedure for the KDQOL-36 (Kidney Disease Quality of Life Instrument adopted for quality of life assessment of patients with kidney disease),first transforms the raw precoded numeric values of items to a 0-100 possible range with higher transformed scores reflecting a better quality of life. Each item is put on a 0 to100 range so that the lowest and highest possible scores are set at 0 and100, respectively. The results entered in the outcome data is the mean absolute difference between the mean pre-test score and the mean post-test score.
Time Frame: 3 month
Population: Subjects were asked to complete a KDQOL-36 (Kidney Disease Quality of Life Instrument adopted for quality of life assessment of patients with kidney disease), once prior to therapy, and then again at the end of 3 months when therapy (when therapy is completed), was completed. Pre and post results will be compared.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Vitamin B12
Number analyzed (Participants) | 57
Scores on a Scale
  Social Function (pre-test) | 56.67 (29.07)
  Social Function (post-test) | 67.50 (24.91)
  Symptom/problem list (pre-test) | 76.62 (18.60)
  Symptom/problem list (post-test) | 75.69 (19.98)
  Effects of kidney disease (pre-test) | 52.29 (26.08)
  Effects of kidney disease (post-test) | 54.58 (26.96)
  Burden of kidney disease pre-test | 43.75 (31.25)
  Burden of kidney disease (post-test) | 37.50 (29.60)
  Work status (pre-test) | 26.67 (32.00)
  Work status (post-test) | 16.67 (30.86)
  Cognitive function (pre-test) | 71.11 (28.91)
  Cognitive function (post-test) | 72.44 (29.26)
  Quality of social interaction (pre-test) | 70.67 (26.04)
  Quality of social interaction (post-test) | 79.11 (18.15)
  Sexual function (pre-test) | 87.50 (17.68)
  Sexual function (post-test) | 100.00 (0.00)
  Sleep (pre-test) | 51.00 (23.81)
  Sleep (post-test) | 51.33 (24.03)
  Social support (pre-test) | 77.78 (32.53)
  Social support (post-test) | 77.78 (29.99)
  Dialysis staff encouragement (pre-test) | 83.33 (15.43)
  Dialysis staff encouragement (post-test) | 82.50 (16.90)
  Overall health (pre-test) | 54.67 (24.46)
  Overall health (post-test) | 60.00 (27.77)
  Patient satisfaction (pre-test) | 71.11 (22.24)
  Patient satisfaction (post-test) | 62.22 (17.21)
  Physical functioning (pre-test) | 39.33 (30.41)
  Physical functioning (post-test) | 37.00 (27.37)
  Role-physical (pre-test) | 28.33 (38.81)
  Role-physical (post-test) | 40.00 (40.97)
  Pain (pre-test) | 55.83 (36.57)
  Pain (post-test) | 65.83 (33.54)
  General health (pre-test) | 36.92 (17.97)
  General health (post-test) | 44.33 (24.56)
  Emotional well-being (pre-test) | 68.00 (21.43)
  Emotional well-being (post-test) | 64.00 (20.51)
  Role-emotional (pre-test) | 35.56 (44.48)
  Role-emotional (post-test) | 55.56 (46.58)
  Energy/fatigue (pre-test) | 40.33 (27.48)
  Energy/fatigue (post-test) | 48.00 (17.61)
  SF-12 physical composite (pre-test) | 34.06 (8.81)
  SF-12 physical composite (post-test) | 36.12 (9.44)
  SF-12 mental composite (pre-test) | 41.88 (11.45)
  SF-12 mental composite (post-test) | 44.83 (11.18)
  Social function (pre to post change) | 10.83 (19.40)
  Symptom/problem list (pre to post change) | -3.13 (14.72)
  Effects of kidney disease (pre to post change) | 2.29 (9.99)
  Burden of kidney disease (pre to post change) | -6.25 (17.52)
  Work status (pre to post change) | -10.00 (20.70)
  Cognitive function (pre to post change) | 1.33 (28.75)
  Quality of social interaction (pre to post change) | 8.44 (25.63)
  Sleep (pre to post change) | 0.33 (20.81)
  Social support (pre to post change) | 0.00 (39.34)
  Dialysis staff encouragement (pre to post change) | -0.83 (21.89)
  Overall health (pre to post change) | 5.33 (19.95)
  Patient satisfaction (pre to post change) | -8.89 (15.26)
  Physical functioning (pre to post change) | -2.33 (17.10)
  Role-physical (pre to post change) | 11.67 (43.16)
  Pain (pre to post change) | 10.00 (36.29)
  General health (pre to post change) | 7.42 (15.81)
  Emotional well-being (pre to post change) | -4.00 (23.71)
  Role-emotional (pre to post change) | 20.00 (46.80)
  Energy/fatigue (pre to post change) | 7.67 (21.29)
  SF-12 physical composite (pre to post change) | 2.06 (8.63)
  SF-12 mental composite (pre to post change) | 2.94 (9.84)
Statistical Analysis 1: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.047, Wilcoxon signed-rank test — P- value for "social function"
Statistical Analysis 2: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.688, Wilcoxon signed-rank test — P- value of " symptom/problem list "
Statistical Analysis 3: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.772, Wilcoxon signed-rank test — P- value of " effects of kidney disease "
Statistical Analysis 4: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.301, Wilcoxon signed-rank test — P-value of " burden of kidney disease "
Statistical Analysis 5: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.250, Wilcoxon signed-rank test — P-value of " work status "
Statistical Analysis 6: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.895, Wilcoxon signed-rank test — P-value of " cognitive function "
Statistical Analysis 7: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.281, Wilcoxon signed-rank test — P-value of " quality of social interaction "
Statistical Analysis 8: Comparison: Vitamin B12; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test — P-value of " sleep "
Statistical Analysis 9: Comparison: Vitamin B12; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test — P-value of " social support "
Statistical Analysis 10: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.943, Wilcoxon signed-rank test — P-value of " dialysis staff encouragement "
Statistical Analysis 11: Comparison: Vitamin B12; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test — P-value of " overall health "
Statistical Analysis 12: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.090, Wilcoxon signed-rank test — P-value of " patient satisfaction "
Statistical Analysis 13: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.391, Wilcoxon signed-rank test — P-value of " physical functioning "
Statistical Analysis 14: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.438, Wilcoxon signed-rank test — P-value of " role-physical "
Statistical Analysis 15: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.424, Wilcoxon signed-rank test — P-value of " pain "
Statistical Analysis 16: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.169, Wilcoxon signed-rank test — P-value of " general health "
Statistical Analysis 17: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.858, Wilcoxon signed-rank test — P-value of " emotional well-being "
Statistical Analysis 18: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.156, Wilcoxon signed-rank test — P-value of " role-emotional "
Statistical Analysis 19: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.084, Wilcoxon signed-rank test — P-value of " energy/fatigue "
Statistical Analysis 20: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.583, Wilcoxon signed-rank test — P-value of " SF-12 physical composite "
Statistical Analysis 21: Comparison: Vitamin B12; Test type: Superiority or Other; p = 0.358, Wilcoxon signed-rank test — p-value of " SF-12 mental composite "

ADVERSE EVENTS:
Arm/Group | Vitamin B12
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

LIMITATIONS AND CAVEATS:
There were too few patients with MMA levels over 800 to determine sensitivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes